CLINICAL TRIAL: NCT05075213
Title: QuitBet Phase II: A Digital Social Game That Pays You to Stop Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WayBetter, Inc. (Industry)
Collaborators: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QuitBet Phase II
Record Dates: First submitted 2021-09-17; First posted 2021-10-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QuitBet (Experimental): QuitBet is a quit smoking game delivered via a smartphone application that lasts 28 days and includes contingency management in the form of a deposit contract, integrated exhaled breath carbon monoxide (CO) testing, a social feed on which "players" can post and respond to messages, and a "leaderboard" that displays players' status (i.e., whether they are still eligible to win). A game host will post educational information about smoking cessation and serve as a discussion moderator. Participants will deposit ("bet") $30 of their own money at the start of the game. Participants who submit a CO test that is 6ppm or lower (indicating no smoking) on at least 24 of the 26 days between day 3-28 will be declared winners and will split the pot of money that was deposited. All participants who submit at least 21 CO tests during the 28 day game, regardless of the CO test result, will be entered into a lottery to win a prize worth $75.
  Interventions: Behavioral: contingency management (deposit contract); Behavioral: leaderboard and social feed
- QuitBet-NS (no social elements) (Active Comparator): QuitBet-NS will include the deposit contract and integrated CO testing with identical rules to QuitBet for being a winner, the $75 raffle for submitting at least 21 CO tests, a display of the participant's daily CO test results that is updated in real time, and a game feed on which only the game host has the ability to post. Players will not be able to post on this feed or respond to the host's posts. At the beginning of the game, the host will post limited information, including a list of smoking cessation resources. QuitBet-NS will NOT include the social feed, leaderboard, or any other social features.
  Interventions: Behavioral: contingency management (deposit contract); Behavioral: smoking cessation resource list

INTERVENTIONS:
Behavioral: contingency management (deposit contract) — Participants will deposit $30 of their own money to play QuitBet. Participants will submit a CO test once per day between the hours of noon and 11:59pm. Participants whose CO test is 6ppm or lower (indicating no smoking) on at least 24 of 26 days between day 3-28 of the game will be declared winners and split the pot of deposited money. Participants who submit at least 21 CO tests, regardless of the result, will be entered into a raffle to win a prize worth $75.
Behavioral: leaderboard and social feed — Participants will have access to a discussion board on which participants can post and respond to messages to each other. Also, a game host will post educational information about smoking cessation and serve as a discussion moderator.
  Arms: QuitBet
Behavioral: smoking cessation resource list — Participants will have access to a list of smoking cessation resources
  Arms: QuitBet-NS (no social elements)

SUMMARY:
This study is a randomized controlled trial (RCT) of QuitBet, a digital contingency management program for smoking cessation. QuitBet combines social gaming elements with participant-funded financial incentives in the form of a deposit contract. QuitBet "players" deposit (called the "bet") a specified amount of their own money into the game's "pot." All "winners" who achieve the game's goal split the pot equally, such that their bet is fully refunded plus they receive extra money from the forfeited bets of players who did not meet the goal. Participants (N = 550) will be randomly assigned to QuitBet or QuitBet-NS (deposit contract only, no social elements). All participants will be offered a second game after their first game (up to 8 weeks total game duration) and will be asked to complete a survey after each game and at 1 and 4 months after the end of the second game (3 and 6 months after the start of their first game). The study will compare QuitBet vs. QuitBet-NS on smoking behavior outcomes and examine potential mediators of outcomes such as motivation, engagement, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient English fluency to complete study procedures
2. At least 21 years of age
3. U.S. resident of any state
4. currently smokes at least 5 cigarettes per day
5. has an email address
6. has a mailing address at which they can receive packages
7. owns an Internet-connected Apple iPhone or Android smartphone that is compatible with QuitBet
8. willing to deposit $30 via PayPal or a credit card
9. willing to receive financial incentives earned during QuitBet via PayPal or in a paper check sent by mail

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence from combustible tobacco use | 6 months follow-up from the start date of their first QuitBet game

SECONDARY OUTCOMES:
proportion of participants who choose to play a second game | 4 weeks after the start date of their first QuitBet game (end of game)
smoking heaviness | 6 months follow-up from the start of their first QuitBet game
  number of cigarettes smoked during the past 7 days
proportion of participants who use smoking cessation medication | 6 months follow-up from the start of their first QuitBet game

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Rosen, Principal Investigator — WayBetter, Inc.
Locations (1):
- WayBetter, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided